CLINICAL TRIAL: NCT05242809
Title: Development and Feasibility Testing of a Group-based PFMT Programme for Antenatal Women in Nanjing City in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Nanjing Maternity and Child Health Care Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20220107
Record Dates: First submitted 2022-01-24; First posted 2022-02-16 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2022-08

CONDITIONS: Urinary Incontinence
Keywords: Urinary Incontinence; Pelvic floor muscle training
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: The participants will be randomly allocated to two arms: intervention group and control group.
Who Masked: Outcomes Assessor
Masking Description: The principal researcher as the outcome assessor will be blinded when analyzing quantitative data, for example, the demographic data and scores of ICIQ-SF, but will not be blinded to the qualitative interview data, as these interviews will be conducted by the principal researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group receives standard care, which means the participants will receive verbal instruction on PFMT from midwives without any further supervision. For reasons of equipoise, women in the comparator group will be offered the group-based PFMT intervention at the end of the study if they wish.
- Group-based PFMT group (Experimental): The participants in the intervention group will receive PFMT supervision in groups. The number of women per group and the detail of the intervention will be decided through stakeholder development group meetings.The intervention will be teaching the participants to do PFMT in groups. The intervention will help women to identify their pelvic floor muscles and then guide them how to contract the pelvic floor muscle correctly (the detail of the intervention will be discussed and determined in phase 1 of this project).
  Interventions: Behavioral: Group-based PFMT group

INTERVENTIONS:
Behavioral: Group-based PFMT group — The intervention group receives PFMT supervision in groups of about 6-8 women
  Arms: Group-based PFMT group

SUMMARY:
The main objective is to co-design and assess the practicality of group-based Pelvic floor muscle training (PFMT) programme in pregnant women. The co-design of the PFMT programme will involve the stakeholder meeting. The feasibility of the group-based Pelvic floor muscle training (PFMT) programme will be achieved by using ICIQ-SF questionnaire before intervention, the completion time of the intervention and 42-day after delivery. Pregnant women with or without UI at Nanjing maternity and child health care hospital will be offered to participate if they meet the criteria of the research. Participants will be randomized into two groups, interventions and control group that gets standard care at the hospital. The intervention group will meet the midwife to receive supervised group-based PFMT once a month for 4 months in groups. Doing correct PFMT during pregnancy can help women to prevent or decrease the risk of developing UI in pregnancy and postnatal period.

DETAILED DESCRIPTION:
This study is to co-design and assess the practicality of group-based Pelvic floor muscle training (PFMT) programme in pregnant women.

PFMT has been recommended as the first-line treatment for stress urinary incontinence and the other types of urinary incontinence (UI), however, it was not well implemented in many countries due the lack of human resource and financial support. Compared to individual PFMT supervision, which is commonly conducted in hospital with additional fees, delivering PFMT in groups can help more women. Therefore, this study is to codesign and investigate the feasibility of group-based PFMT programme.

The first phase is to co-design the group-based PFMT programme: The stakeholders will be involved in this phase. The stakeholder development group will purposively sample both health professionals and pregnant women with or without UI. The stakeholder development group members will include the principal researcher, two pregnant women without UI, two pregnant women with a history of UI, two midwives (one of the midwives will help the principal researcher to deliver the training session), two physiotherapists. Data from group meetings will be digitally audio-recorded following consent and notes will be taken during the meeting. The data will be analyzed to identify the content and mode of delivery of the group-based PFMT programme along with potential barriers and facilitators.

The second phase is implementation and evaluation of the group-based PFMT programme (randomised controlled feasibility study): Participants will be randomized into two groups, intervention and control group. The control group gets standard care at the hospital. The interventional group gets supervised group-based PFMT. The intervention will be teaching the participants to do PFMT in groups. The intervention will help women to identify their pelvic floor muscles and then guide them how to contract the pelvic floor muscle correctly (the detail of the intervention will be discussed and determined in phase 1 of this project). The core outcome measures are likely to include self-reported UI, which is commonly used in studies and is able to evaluate the effectiveness of PFMT intervention in pregnant women, and UI severity which may be assessed by ICIQ-SF (a validated questionnaire which both assesses the severity of urinary loss and quality of life impact). The adherence to the programme may be assessed by attendance records from the group-based training sessions and completion of a training diary which includes the frequency and duration the participants self-report doing the exercises. The training diary will be submitted to the principal researcher after the training sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Nulliparous women who are aged 18 years and older;
2. Gestational ages of 19-24 weeks;
3. With or without the symptom of UI;
4. Singleton fetus
5. Capable of giving valid informed consent

Exclusion Criteria:

1. Women with pregnancy complications or urine tract infection
2. Women with previous UI symptoms before pregnancy
3. High risk of preterm labour
4. Women with previous urogenital surgery or diseases which may interfere with pelvic floor muscle strength, for example, pelvic organ prolapse, neurological disorders, diabetes.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-08-21 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
self-reported UI change | baseline(before the intervention starts, week 0); completion of the intervention (week 13); 42 days after delivery (an average of week 19 to week 20)
  assessed by International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF). The third question in this questionnaire is the frequency of UI which can present the self-reported UI change.
the impact of UI on quality of life change | baseline(before the intervention starts, week 0); completion of the intervention (week 13); 42 days after delivery (an average of week 19 to week 20)
  assessed by International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF). The fifth question is the overall impact of UI which ranged from 0 to 10. In the scale, 0 means the impact on life is not at all while 10 means the impact on life is a great deal with larger number represents greater impact on life.
adherence to PFMT programme change 1 | completion of the intervention (week 13)
  assessed by attendance records from the group-based training sessions
adherence to PFMT programme change 2 | completion of the intervention (week 13)
  assessed by record of a training diary which includes the frequency the participants self-report doing the exercises.

SECONDARY OUTCOMES:
Recruitment rates | completion of the intervention (week 13)
  The percentage of participants take part in the intervention
Retention of participants | completion of the intervention (week 13)
  The percentage of participants who complete the intervention
The acceptability of randomization | completion of the intervention (week 13)
  This is a qualitative measure which will be assessed through semi-structured interview. The participants will be asked whether randomization is acceptable and the reason if the answer is not.
The acceptability of the outcome measures | completion of the intervention (week 13)
  This is a qualitative measure which will be assessed through semi-structured interview. The participants will be asked whether the outcome measures are acceptable and the reason if the answer is not.
The completion rates of the outcome measures | completion of the intervention (week 13)
  The percentage of the participants complete the ICIQ-SF and the training diary.
participants' advice on group-based PFMT programme | completion of the intervention (week 13)
  This is a qualitative measure which will be assessed through semi-structured interview.
midwife's advice on group-based PFMT programme | completion of the intervention (week 13)
  This is a qualitative measure which will be assessed through semi-structured interview.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Maternity and Child Health Care Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang X, Zhang A, Sayer L, Bassett S, Woodward S. Co-design of a group-based programme to facilitate adherence to pelvic floor muscle training in pregnant women in China: Describing the process of developing an intervention underpinned by the behaviour change wheel. Midwifery. 2025 May;144:104316. doi: 10.1016/j.midw.2025.104316. Epub 2025 Feb 10. PMID 40037186
- [Derived] Yang X, Sayer L, Bassett S, Woodward S. Group-based pelvic floor muscle training for pregnant women: A randomized controlled feasibility study. J Adv Nurs. 2025 Apr;81(4):2099-2112. doi: 10.1111/jan.16365. Epub 2024 Aug 14. PMID 39140698
- [Derived] Yang X, Zhang A, Zhu R, Sayer L, Bassett S, Woodward S. Group-based PFMT programme for preventing and/or treating UI in pregnant women: protocol of a randomized controlled feasibility study. Pilot Feasibility Stud. 2023 Oct 31;9(1):180. doi: 10.1186/s40814-023-01410-2. PMID 37907990